CLINICAL TRIAL: NCT04762550
Title: Diagnosis and Management of Impaired Thrombin Generation in Liver Transplant Surgery
Brief Title: Thrombin Generation in Liver Transplant Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5414.0
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-02

CONDITIONS: Liver Transplantation; Thrombin; Hemostasis, Surgical; Blood Coagulation Disorder Due to Liver Disease; Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma specimens in citrated tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Liver Transplantation: This is a prospective observational study that intends to offer participation to all patients undergoing liver transplantation at Toronto General Hospital. Parameters that will be measured include Thrombin generation, viscoelastic testing utilizing ROTEM, and conventional laboratory testing (INR, aPTT and Fibrinogen level) at five time points: (a) Prior to cross-clamp application; (b) within the first 30 minutes of venous cross clamp removal; (c) after 30 minutes of reperfusion; (d) On arrival in the intensive care unit (ICU) or post-anesthesia recovery unit; and (5) 12 hours post-operatively.

SUMMARY:
This is a prospective observational study of 100 patients undergoing liver transplantation at a single centre. Thrombin generation and kinetics will be assessed using a novel point-of-care device, and compared to conventional measures of hemostasis as well as viscoelastic tests to pinpoint specific coagulation deficits and identify potential therapeutic targets. The clinical course of patients will be followed for major bleeding and transfusion outcomes.

DETAILED DESCRIPTION:
Liver transplantation is the only curative option for end stage liver disease, but is associated with high morbidity and mortality. End stage liver disease is known to be accompanied by dysregulated coagulation, which is further exacerbated in the immediate perioperative period by transplantation, leading to both coagulopathic bleeding and thrombosis. Altered thrombin generation is thought to play a key role in the predisposition of these patients for both severe coagulopathic hemorrhage and life-threatening thromboembolic complications. Despite this, thrombin generation during the immediate transplant period in patients with end-stage liver disease is poorly characterized, in part because it is not well reflected by conventional measures of coagulation. This study aims to characterize changes in thrombin generation capacity pre, intra- and post-transplant utilizing a novel point-of-care thrombin generation assay. Other specific aims of the study are to identify risk factors for patients with impaired thrombin generation and will assess the association of impaired thrombin generation with overall clinical bleeding risk. The overarching goal of this work is to develop a point-of-care-testing guided algorithm addressing dysregulated thrombin formation that improves coagulation management without increasing the risk of thromboembolic complications. Ultimately, this line of research will improve the outcomes of liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (> 18 years of age) proceeding to imminent (within 24 hours) liver transplantation surgery at Toronto General Hospital will be offered participation.
* Patients should have end stage liver disease necessitating transplantation. All etiologies of end stage liver disease will be accepted.

Exclusion Criteria:

- Patients who are unable to consent to the study or who refuse participation will be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consenting adults undergoing liver transplantation surgery at Toronto General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Thrombin Generation - Endogenous Thrombin Potential (nM*min) | The pattern of change in thrombin generation will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The change in thrombin generation will be measured in patients undergoing liver transplantation, as assessed through the Endogenous Thrombin Potential (nM*min)
Thrombin Generation - Lag Time (Seconds) | The pattern of change in thrombin generation will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The change in thrombin generation will be measured in patients undergoing liver transplantation as assessed by the Lag Time (Seconds)
Thrombin Generation - Time to Peak (Seconds) | The pattern of change in thrombin generation will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The change in thrombin generation will be measured in patients undergoing liver transplantation by the Time to Peak (Seconds)
Thrombin Generation - Peak Height (nM) | The pattern of change in thrombin generation will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The change in thrombin generation will be measured in patients undergoing liver transplantation by the Peak Height (nM)

SECONDARY OUTCOMES:
Conventional Hemostatic Tests - Platelet Count | The pattern of change will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The platelet count from the complete blood count in x10^9/L
Conventional Hemostatic Tests - INR | The pattern of change will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The international normalized ratio (INR) in seconds
Conventional Hemostatic Tests - aPTT | The pattern of change will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The activated partial thromboplastin time (aPTT) in seconds
Conventional Hemostatic Tests - Fibrinogen Level | The pattern of change will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  The Clauss Fibrinogen level in g/L
Viscoelastic Testing | The pattern of change will be assessed intra-operatively at baseline through to study completion up to 12 hours post-operatively
  Rotational thromboelastometry (ROTEM)

OTHER OUTCOMES:
Transfusion Outcomes - Red Blood Cells | From intra-operatively to within 12 hours post-operatively
  The total number of red blood cells transfused
Transfusion Outcomes - Platelets | From intra-operatively to within 12 hours post-operatively
  The total number of platelet units transfused
Transfusion Outcomes - Frozen Plasma | From intra-operatively to within 12 hours post-operatively
  The total number of frozen plasma units transfused
Transfusion Outcomes - Prothrombin Complex Concentrate | From intra-operatively to within 12 hours post-operatively
  The total number of units transfused
Transfusion Outcomes - Fibrinogen Concentrate | From intra-operatively to within 12 hours post-operatively
  The total number of grams of fibrinogen transfused
Bleeding Outcomes - Delayed Abdominal Closure | From intra-operatively to within 12 hours post-operatively
  Clinical bleeding outcome such as delayed abdominal
Bleeding Outcomes - Return to the Operating Room for Re-Exploration | From intra-operatively to within 12 hours post-operatively
  Clinical bleeding outcome such as return to the operating room for re-exploration or evacuation of hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Bartoszko, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network; Keyvan Karkouti, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No